CLINICAL TRIAL: NCT05580653
Title: Phase 1 Seattle Dietary Biomarkers Development Center
Acronym: P1-SDBDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marian Neuhouser (Other)
Collaborators: United States Department of Agriculture - National Institute of Food and Agriculture (USDA-NIFA) (Unknown); University of Nebraska (Other); University of Washington (Other); Duke University (Other)
Responsible Party: Sponsor-Investigator, Marian Neuhouser, Professor, Cancer Prevention Program Head, Fred Hutchinson Cancer Center
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: RG1121654; USDA-NIFA 2022-67017-38475 (Other Grant/Funding Number: United States Department of Agriculture - National Institute of Food and Agriculture (USDA-NIFA))
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy Adults
Keywords: Healthy Diet; Diet; Red meat; Eggs; Pinto beans; Black beans; Pharmacokinetics; Metabolomics

STUDY DESIGN:
Intervention Model Description: Randomized cross-over
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statisticians, Laboratory personnel
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 1) Beef then half beef and half pinto bean then pinto bean (Experimental)
  Interventions: Other: Controlled feeding study of beef and/or pinto beans
- 2) Half pinto bean and half beef then pinto bean then beef (Experimental)
  Interventions: Other: Controlled feeding study of beef and/or pinto beans
- 3) Pinto Bean then Beef then half pinto bean and half beef (Experimental)
  Interventions: Other: Controlled feeding study of beef and/or pinto beans
- 4) Egg then half Egg and half black bean then black bean (Experimental)
  Interventions: Other: Controlled feeding study of eggs and/or black beans
- 5) Half egg and half black bean, then black bean then egg (Experimental)
  Interventions: Other: Controlled feeding study of eggs and/or black beans
- 6) Black bean then egg then half black bean and half egg (Experimental)
  Interventions: Other: Controlled feeding study of eggs and/or black beans

INTERVENTIONS:
Other: Controlled feeding study of beef and/or pinto beans — Crossover feeding study of three, 7-day feeding periods with plant and/or animal proteins (beef, pinto beans, and half beef/half pinto beans) completed in random order.
  Arms: 1) Beef then half beef and half pinto bean then pinto bean; 2) Half pinto bean and half beef then pinto bean then beef; 3) Pinto Bean then Beef then half pinto bean and half beef
Other: Controlled feeding study of eggs and/or black beans — Crossover feeding study of three, 7-day feeding periods with plant and/or animal proteins (eggs, black beans, and half eggs/half black beans) completed in random order.
  Arms: 4) Egg then half Egg and half black bean then black bean; 5) Half egg and half black bean, then black bean then egg; 6) Black bean then egg then half black bean and half egg

SUMMARY:
The Seattle Dietary Biomarker Development Center (S-DBDC) aims to advance the science of measuring dietary intake by identification and validation of dietary biomarkers that improve upon self-reported diet. To accomplish this mission, the Seattle DBDC will carry out controlled feeding studies in healthy human volunteers. Metabolomics assays will be conducted on blood and urine specimens collected during the feeding studies for biomarker identification.

DETAILED DESCRIPTION:
The central mission of the Seattle Dietary Biomarker Development (DBDC) is to advance the science of measuring complex dietary exposures by rigorous identification and validation of dietary biomarkers that improve upon measurement error prone self-reported diet. To accomplish this mission, the Seattle DBDC will conduct a set of two, randomized, crossover, 3-period controlled feeding trials to develop metabolomics-based blood and urine biomarkers of 4 individual foods (1) beef and pinto beans or 2) eggs and black beans) and determine the dynamic ranges and half-lives of the urinary and blood-based dietary biomarkers. The two trials use the exact same sample protocol and study procedures and will be conducted successively.

For each feeding trial, 15 healthy adults will complete three feeding periods in random order (all protein from beef (trial 1) or eggs (trial 2); 1/2 protein from beef (trial 1) or eggs (trial 2); and 1/2 protein from pinto beans (trial 1) or black beans (trial 2); all protein from pinto beans (trial 1) or black beans (trial 2)). Each feeding period will consist of a 2-day run-in of controlled feeding followed by a 7-day feeding period, with about a 7-day washout between feeding periods. Blood and urine specimens will be collected before, at the mid-point, and at the end of each feeding period. In addition, an all-day pharmacokinetic evaluation will be conducted for 2 of the 3 feeding periods (all beef and all pinto beans (trial 1); all eggs and all black beans (trial 2)). Stool samples will be collected before, and at the end of each feeding period and stored for future studies. The collected specimens will be used for study outcomes and archived for future studies.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults
2. Age 18 years and older
3. Willing to come to the Fred Hutch campus 16 times during the study
4. BMI 18.5-39.9 kg/m2

Exclusion Criteria:

1. History of gastrointestinal disorders (e.g., ulcerative colitis, Crohn disease, celiac sprue, Hereditary Non-polyposis Colorectal Cancer, familial adenomatous polyposis, pancreatic disease, liver disease)
2. Bleeding disorder that precludes blood draws
3. Previous gastrointestinal resection or bariatric surgery
4. Recent hospital admissions (in past 6 months) for heart disease (myocardial Infarction/cerebrovascular accident or congestive heart failure) or other cardiovascular disease/coronary artery disease condition under physician guided therapy that is not medically stable.
5. Cancer under active radiation or chemotherapy treatment (post-6 mos)
6. Pregnant or lactating
7. Weight change (±5% in 3 months)
8. Regular alcohol intake of >2 drinks/day (2 drinks being equivalent to 720 ml beer, 240 ml wine, or 90 ml spirits) and unwilling to abstain during feeding periods
9. Use of tobacco and/or marijuana, hookahs, e-cigarettes (e-cigs, vaping devices, etc) and not willing to abstain during feeding periods.
10. Use of illicit drugs and not willing to abstain during feeding periods.
11. BMI ≥40 kg/m2
12. Seated blood pressure > 140/90 mm Hg
13. Fasting clinical lab tests outside acceptable value as ascertained at a screening blood draw°
14. Food allergies/intolerances or major dislikes to foods used in the study menus; unwilling to consume study foods.
15. Current use of specific prescription medication (study staff will review medications to determine eligibility)**
16. Regular (daily to weekly) use of over-the-counter weight-loss aids, anti-inflammatories, and unable to stop taking these during feeding periods
17. Unwilling to stop taking OTC dietary supplements that interfere with the test foods being studied, including pills, chewables, liquids or powders for the following: protein supplements, soy, fiber, flaxseed, fish oil (incl. cod liver oil), probiotics, glucosamine and chondroitin (if vitamin supplement is MD prescribed - may continue). Study staff will review supplements to determine eligibility
18. Oral or IV antibiotic use in the past 3 months (could defer participation until 3 months post completion of course of antibiotics)
19. Inability to freely give informed consent.

    * Fasting clinical lab tests outside acceptable value as ascertained at a screening blood draw:

Description [Acceptable Values]

Glucose-Fasting: Serum Glucose [54-125 mg/dl]

Urea: BUN [6-50mg/dl]

Serum Creatinine [0.4-1.3 mg/dl]

eGFR: estimated GFR [>60ml/min]

Serum Sodium [133-146 mmol/L]

ALT/GPT Liver Enzyme [5-60 U/L]

AST/GOT Liver Enzyme [5-40 U/L]

Alkaline Phosphatase Liver Enzyme [20-135 U/L]

Total Bilirubin Liver Function [0.0-1.9 mg/dl]

Total Serum Protein [5-9.0 g/dl]

Albumin Serum Protein [3.5-5.9 g/dl]

LDL Cholesterol [<160 mg/dl]

Triglycerides [<500 mg/dl]

WBC White Blood Cells [3-10.5 K/uL]

HCT (women) Hematocrit [35-48 g/dl]

HCT (men) Hematocrit [37.5-49 g/dl]

**Medication use for exclusion:

1. Diuretics
2. Steroids (oral): daily oral any dose within 1 month of study, except OCP as noted below
3. Opiates: any use within 1 month of study
4. Anti-lipid medications that affect GI or renal function (ie. Fibrates)
5. Hyperglycemia medications other than metformin (ie. insulin, SGLT2 inhibitor, α-glucosidase inhibitor)
6. Psychiatric that affect metabolism/renal function (anti-psychotics, lithium)
7. Biologic/immune modulators (ie. RA, psoriasis, other rheumatologic/hematologic active disease)
8. Anti-coagulants (coumadin, heparin, Eliquis, etc.)
9. HIV/HAART, etc. (dyslipidemic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Mean metabolite concentration at Day 7 for Beef | Day 7
Mean metabolite concentration at Day 7 for Pinto Bean | Day 7
Mean area under the curve of 24-hour metabolite concentration for Beef | 0-24 hours
Mean area under the curve of 24-hour metabolite concentration for Pinto Bean | 0-24 hours
Mean metabolite concentration at Day 7 for Egg | Day 7
Mean metabolite concentration at Day 7 for Black Bean | Day 7
Mean area under the curve of 24-hour metabolite concentration for Egg | 0-24 hours
Mean area under the curve of 24-hour metabolite concentration for Black Bean | 0-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marian L. Neuhouser, PhD, RD, Principal Investigator — Fred Hutchinson Cancer Center; Johanna W. Lampe, PhD, RD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We will comply with the NIH Data Sharing Policy. This trial will be registered at ClinicalTrials.gov. We will publish results in peer-reviewed journals. Data generated from this study will be sent to the Data Coordinating Center Center (DCC) at Duke University. The DCC will make study data available to other Consortium members (University of California Davis, Harvard University) in accordance with best practices for data safety and accessibility. Participants' data may be stored and shared for future research without additional informed consent if identifiable private information is removed. Use of participant data may result in commercial profit; however, participants will not be compensated for the use of their data other than what is described in the consent form. The final de-identified study data and results will be made publicly available, in accordance with NIH data sharing policies.
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Chakraborty H, Sun Q, Bhupathiraju SN, Schenk JM, Mishchuk DO, Bain JR, He X, Sun J, Harnly J, Simmons W, Raftery D, Liang L, Newman JW, Fiehn O, Clish CB, Lampe JW, Bennett BJ, Navarro SL, Wang Y, Zheng C, Mossavar-Rahmani Y, McCullough ML, Huang Y, Shojaie A, Zhu W, Djukovic D, Sacks F, Williams J, Steinberg FM, Adams SH, Hu FB, Neuhouser ML, Slupsky CM, Maruvada P. The Dietary Biomarkers Development Consortium: An Initiative for Discovery and Validation of Dietary Biomarkers for Precision Nutrition. Curr Dev Nutr. 2025 Apr 5;9(5):107435. doi: 10.1016/j.cdnut.2025.107435. eCollection 2025 May. PMID 40641655

DOCUMENTS (2):
  • Informed Consent Form: Beef version (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT05580653/ICF_000.pdf
  • Informed Consent Form: Egg version (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/53/NCT05580653/ICF_001.pdf